CLINICAL TRIAL: NCT05347017
Title: The Effect of Autogenous Demineralized Dentin Block Graft Versus Autogenous Bone Block Graft on Alveolar Ridge Preservation: A Randomized Controlled Clinical Trial
Brief Title: Autogenous Demineralized Dentin Block Graft Versus Autogenous Bone Block Graft for Alveolar Ridge Preservation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Talaat Mohamed Mahmoud El Behwashy, Principal Investigator. Mohamed Elbehwashy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: perio2022april
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alveolar ridge preservation using autogenous demineralized dentin block graft (Experimental): Atraumatic extraction of non-restorable teeth, then the extracted tooth will be prepared and demineralized using HCL acid as demineralized dentin block graft and inserted in the extraction socket
  Interventions: Procedure: Alveolar ridge preservation using autogenous demineralized dentin block graft
- Alveolar ridge preservation using autogenous bone block graft (Active Comparator): Atraumatic extraction of non-restorable teeth, then autogenous bone block will be harvested from the maxillary tuberosity and reshaped and inserted in the extraction socket
  Interventions: Procedure: Alveolar ridge preservation using autogenous bone block graft

INTERVENTIONS:
Procedure: Alveolar ridge preservation using autogenous demineralized dentin block graft — Atraumatic extraction of non restorable tooth, then the extracted tooth will be prepared and demineralized by HCL acid and inserted as demineralized dentin block graft in the socket
  Arms: Alveolar ridge preservation using autogenous demineralized dentin block graft
Procedure: Alveolar ridge preservation using autogenous bone block graft — Atraumatic extraction of non restorable tooth, then the autogenous bone block graft will be harvested from the maxillary tuberosity and reshaped and inserted into the socket
  Arms: Alveolar ridge preservation using autogenous bone block graft

SUMMARY:
The aim of this trial is to compare the effect of autogenous demineralized dentin block graft (ADDBG) versus autogenous bone block graft (ABBG) harvested from maxillary tuberosity on alveolar ridge preservation after extraction of non-restorable single rooted teeth

DETAILED DESCRIPTION:
Many studies have reported an approximately 50% reduction in alveolar bone both the horizontal and vertical directions over 12 months with more than two-thirds of the reduction occurring in the first three months after extraction. Alveolar ridge preservation is a procedure that attempts to reduce bone dimensional changes that naturally take place following tooth extraction. A broadly recognized approach is the maintenance of bone walls through bone substitute (graft) delivery into the socket, where guided bone regeneration may be a requisite. Autogenous bone graft has osteogenic and osteoinductive effect. however, when attempts were made to use autologous bone chips in socket preservation, they failed to promote healing or stimulate hard tissue formation in the socket. On the other hand, autogenous bone block graft from the tuberosity has shown a feasible, user-friendly, low-cost solution for minimizing soft and hard tissue collapse and dimensional loss following single-rooted tooth extraction.

Moreover, root dentin block is composed of Type I collagen matrix with several osteoinductive non-collagenous proteins such as bone morphogenetic proteins (BMP) and dentin matrix proteins. Geometrically, alveolar bone morphology was maintained by dentin block graft as well as it has micropores (dentinal tubules) of 3-5 μm diameter and macropores of 0.2-0.3 mm diameter for enhancing osteoinductive and osteoconductive functions.

Both demineralized dentin block and autogenous bone block grafts has been utilized for alveolar ridge preservation or augmentation but the superiority of one form over the other is not yet clear

ELIGIBILITY:
Inclusion Criteria:

* Non-restorable tooth indicated for extraction
* Single-rooted teeth
* Motivated patients, agree to sign informed consent and complete the follow-up period

Exclusion Criteria:

* Pregnant females
* active infection at extraction site
* Smokers
* systemic conditions affecting healing (e.g. diabetes, medications as bisphosphonates...)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Alveolar ridge bucco-lingual width change in mm | 6 months
  Alveolar bone linear width will be measured at baseline and after 6 months using cone beam computed tomography (CBCT) scans. The change in bone width will be calculated as the subtraction of final width from baseline width and will be measured in millimetres (Jung et al., 2013)

SECONDARY OUTCOMES:
Alveolar ridge apico-coronal height change in mm | 6 months
  Difference in height linear measurement between baseline and final CBCT scans (Jung et al., 2013)
  Difference in height linear measurement between baseline and final CBCT scans (Jung et al., 2013)
  Measures the difference in height linear measurements between baseline and final CBCT scans (Jung et al., 2013)
Histological assessment | 6 months
  Bone samples from control and intervention sites will be taken during implant placement using a trephine bur of a size smaller than the implant. Samples will be examined for new bone formation (Yes/no) and inflammatory response (Yes/no) (Wong and Rabie, 2010).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jung RE, Philipp A, Annen BM, Signorelli L, Thoma DS, Hammerle CH, Attin T, Schmidlin P. Radiographic evaluation of different techniques for ridge preservation after tooth extraction: a randomized controlled clinical trial. J Clin Periodontol. 2013 Jan;40(1):90-8. doi: 10.1111/jcpe.12027. Epub 2012 Nov 19. PMID 23163915
- [Background] Wong RW, Rabie AB. Effect of bio-oss collagen and collagen matrix on bone formation. Open Biomed Eng J. 2010 Mar 9;4:71-6. doi: 10.2174/1874120701004010071. PMID 20461225
- [Background] Barootchi S, Wang HL, Ravida A, Ben Amor F, Riccitiello F, Rengo C, Paz A, Laino L, Marenzi G, Gasparro R, Sammartino G. Ridge preservation techniques to avoid invasive bone reconstruction: A systematic review and meta-analysis: Naples Consensus Report Working Group C. Int J Oral Implantol (Berl). 2019;12(4):399-416. PMID 31781696
- [Background] Younes R, Khairallah CM. The "One Piece" Autologous Tuberosity Graft: A Contemporary Concept in Ridge Preservation. Case Rep Dent. 2020 Feb 13;2020:3945076. doi: 10.1155/2020/3945076. eCollection 2020. PMID 32099685
- [Background] Kim, Y., Fajardo, K., Valera, A. and Um, I. (2017) 'Autogenous Tooth Bone Graft Block For Socket Preservation: A One-Stage Technique', Dentistry, 7(414), pp. 2161-1122.1000414.